CLINICAL TRIAL: NCT06422156
Title: A Prospective, Multicenter, Single Arm Study of SBRT Combined With Nimotuzumab and Mono-chemotherapy in the Treatment of Locally Advanced Pancreatic Cancer
Brief Title: SBRT Combined With Nimotuzumab and Mono-chemotherapy in Locally Advanced Pancreatic Cancer
Acronym: Nim-PC-28
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Peking University Third Hospital (Other)
Collaborators: Biotech Pharmaceutical Co., Ltd. (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: M2023639
Record Dates: First submitted 2024-03-17; First posted 2024-05-20 (Actual); Last update posted 2024-05-20 (Actual); Status verified 2023-11

CONDITIONS: Advanced Pancreatic Cancer
Keywords: advanced pancreatic cancer; stereotactic body radiation therapy (SBRT); Nimotuzumab
MeSH Terms: interventions — Radiosurgery; nimotuzumab; Drug Therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- SBRT+Nimotuzumab+ mono-chemotherapy (Experimental): All eligible patients will receive SBRT combined with nimotuzumab and mono-chemotherapy.
  Interventions: Radiation: Stereotactic body radiation; Drug: Nimotuzumab; Drug: mono-chemotherapy

INTERVENTIONS:
Radiation: Stereotactic body radiation — Patients will receive SBRT with doses ranging from 35-40 Gy in five fractions.
  Other Names: SBRT
Drug: Nimotuzumab — Patients will receive Nimotuzumab 400 mg weekly or Nimotuzumab 600mg on day 1 and 8 of a 21-day cycle until disease progression.
  Other Names: h-R3
Drug: mono-chemotherapy — Patients will receive mono-chemotherapy (Gemcitabine, S-1 or capecitabine) until disease progression.
  Other Names: chemotherapy

SUMMARY:
This is a prospective, multicenter, single arm clinical study. The main purpose of the study is to evaluate the clinical efficacy and safety of SBRT combined with Nimotuzumab and mono-chemotherapy in the treatment of locally advanced pancreatic cancer (LAPC).

DETAILED DESCRIPTION:
This clinical study is designed as a prospective, multicenter, single arm study to evaluate the clinical efficacy and safety of SBRT combined with nimotuzumab and mono-chemotherapy in the treatment of locally advanced pancreatic cancer (LAPC). All eligible patients will receive SBRT with doses ranging from 35-40 Gy in five fractions, intravenous nimotuzumab 400mg weekly or 600mg on day 1 and 8 of a 21-day cycle, and mono-chemotherapy (Gemcitabine, S-1 or capecitabine) until disease progression, death, unacceptable toxicity, or consent withdrawal. The main endpoint is progression-free survival (PFS).

ELIGIBILITY:
Inclusion Criteria:

* 1. Age 18-75 years old, gender unlimited;
* 2. Histologically or cytologically confirmed pancreatic ductal adenocarcinoma (PDAC);
* 3. Locally advanced pancreatic cancer (according to the NCCN criteria), unresectable or surgically declined;
* 4. The maximum diameter of the primary tumor was < 5.0cm;
* 5. Eastern Cooperative Oncology Group (ECOG) performance status of 0 or 1;
* 6. No prior radiotherapy (upper abdomen) or tumor systemic therapy;
* 7. Adequate organ and bone marrow function, defined as follows: absolute neutrophil count (ANC)≥1.5×10^9/L; hemoglobin≥9.0 g/dL; platelets≥75×10^9/L; serum total bilirubin (TBIL)≤1.5×ULN; aspartate aminotransferase (AST) and alanine aminotransferase (ALT) ≤ 2.5 times the upper limit of normal (ULN); serum creatinine≤1.5×ULN;
* 8. Left ventricular ejection fraction ≥50%;
* 9. Fertile subjects are willing to take contraceptive measures during the study period;
* 10. Woman who are breastfeeding during the study period or within 150 days after the last treatment;
* 11. Survival was expected to be ≥3 months;
* 12.Good compliance and signed informed consent voluntarily.

Exclusion Criteria:

* 1. Tumor invasion of gastrointestinal tract;
* 2. Woman who are pregnant or breastfeeding;
* 3. History of other malignancies (except cured basal cell carcinoma of the skin and carcinoma in situ of the cervix) within the past 5 years;
* 4. History of uncontrolled epilepsy, central nervous system disease, or mental disorder, which may influence the signing of informed consent or affect the patient's adherence;
* 5.Serious heart disease, such as symptomatic coronary heart disease, New York Heart Association (NYHA) class II or more, severe congestive heart failure or severe arrhythmia requiring medical intervention, or a history of myocardial infarction within the past 12 months;
* 6. Patients requiring immunosuppressive;
* 7.Accompanied by active infections, or a major hematological, renal, metabolic, gastrointestinal, endocrine, or metabolic disorder determined by the investigator, or other serious uncontrolled concomitant disease;
* 8. Known allergy to prescription or any component of the prescription used in this study;
* 9. Immunodeficiency, including HIV infection or other acquired immunodeficiency, or a history of organ transplantation, or other immune-related disorders requiring medical intervention;
* 10. Patients with acute and chronic tuberculosis infection;
* 11. Received Chinese herbal medicines or immune-modulators for anti-tumor within 2 weeks prior to initial administration;
* 12.History of noninfectious pneumonia requiring glucocorticoid therapy or current interstitial lung disease within 1 year prior to initial administration;
* 13. Received any other form of immunosuppressive therapy within 7 days prior to the initial of study administration;
* 14. Participated in other clinical trials within 4 weeks, or received another investigational drugs or investigational device within 4 weeks prior to the initial administration;
* 15.Other reasons that are not suitable to participate in this study according to the researcher's judgment.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 73 (Estimated)
Dates: Start 2024-06-01 (Estimated); Primary Completion 2026-06-01 (Estimated); Study Completion 2026-06-01 (Estimated)

PRIMARY OUTCOMES:
progression-free survival (PFS) | Up to 12 months
  PFS, defined as the time from the beginning of treatment to disease progression or all-cause death. Progression is defined using Response Evaluation Criteria In Solid Tumors Criteria (RECIST v1.1), as a 20% increase in the sum of the longest diameter of target lesions, or a measurable increase in a non-target lesion, or the appearance of new lesions.

SECONDARY OUTCOMES:
overall survival (OS) | Up to 12 months
  The time from the beginning of treatment to death due to any cause.
Objective response rate (ORR) | Up to 12 months
  Objective response rate (ORR), including complete response (CR) and partial response (PR). Per Response Evaluation Criteria In Solid Tumors Criteria (RECIST v1.1) for target lesions and assessed by CT/MRI: Complete Response (CR), Disappearance of all target lesions; Partial Response (PR), at least a 30% decrease in the sum of the longest diameter of target lesions.
Disease control rate (DCR) | Up to 12 months
  Disease control rate (DCR), including complete response (CR) and partial response (PR) and stable disease(SD). Per Response Evaluation Criteria In Solid Tumors Criteria (RECIST v1.1) for target lesions and assessed by CT/MRI: CR, disappearance of all target lesions; PR, at least a 30% decrease in the sum of the longest diameter of target lesions. SD, neither sufficient shrinkage to qualify for PR nor sufficient increase to qualify for PD (PD, defined as a 20% increase in the sum of the longest diameter of target lesions, or a measurable increase in a non-target lesion, or the appearance of new lesions).
Pain relief rate | Up to 12 months
  The proportion of patients with pain relief after treatment to the total number enrolled.
adverse events | Up to 30 days after last administration
  Frequency and severity of adverse events.

CONTACTS AND LOCATIONS:
Overall Officials: Junjie Wang, Dr, Principal Investigator — Peking University Third Hospital

IPD SHARING:
Plan to Share IPD: No